CLINICAL TRIAL: NCT06008587
Title: Contribution of Nasal High Flow in Pneumology Assessed in Acid-Free Hypercapnic Acute Respiratory Failure
Acronym: PIRAHNA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossible to achieve inclusion goals, fewer patients in reality than expected
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-CHITS-012; 2022-A02641-42 (Other: ID-RCB number)
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Insufficiency
Keywords: Nasal High Flow; Acute Respiratory Failure; Respiratory non-acidosis; Pneumology; Hypercapnia
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal High Flow therapy in association with the standard therapy (Experimental)
  Interventions: Device: AIRVO3 TM; Other: Standard therapy
- Standard therapy alone (Active Comparator)
  Interventions: Other: Standard therapy

INTERVENTIONS:
Device: AIRVO3 TM — A device that provides high flows of heated and humidified respiratory gases to patient who breath spontaneously. Patients will be treated with the device up to 15 days or until the occurrence of respiratory acidosis defined by pH<7.35, whichever come first.
  Arms: Nasal High Flow therapy in association with the standard therapy
Other: Standard therapy — Standard therapy depends on the acute respiratory failure etiology. Treatments will be administered at the investigator's discretion in accordance with the standard of care.

SUMMARY:
The hypothesis is that Nasal High Flow therapy for patients with Hypercapnic Acute Respiratory Failure without acidosis, in addition to standard treatment would improve the care.

DETAILED DESCRIPTION:
The aim of the PIRAHNA study is to compare patients treated with Nasal High Flow in association with conventional standard treatment versus patients treated only with conventional standard treatment.

Primary objective : To demonstrate the therapeutic superiority of Nasal High Flow in hypercapnic Acute Respiratory Failure without acidosis, in combination with conventional standard treatment

Secondary objectives :

1. Identify the characteristics (etiologies) of responder patients (defined by a decrease in capnia and a failure to develop acidosis within two weeks of hospitalization)
2. Identify the etiology (trigger) of the Acute Respiratory Failure of responder patients
3. Compare the evolution of respiratory rate between the two treatment groups
4. Compare the evolution of dyspnea between the two treatment groups
5. Compare the evolution of gas exchanges between the two treatment groups
6. Compare the length of stay between the two groups
7. Compare the evolution of patients comfort state in the two treatment groups

ELIGIBILITY:
Inclusion Criteria:

* Major patient ≥ 18 years old
* Medical diagnosis of Acute Respiratory Failure less than 48 hours
* With partial pressure of carbon dioxide (PaCO2) > 45 and pH > 7.35 for less than 48 hours, with no indication of Non-Invasive Ventilation (NIV) placement
* Underlying terrain of known or unknown chronic respiratory pathology (may be unknown at time of diagnosis) Examples : COPD, Bronchiectasis, Pulmonary fibrosis, asthma, sequelae pathologies …
* All etiologies (infectious, cardiac decompensation, trauma, etc.)
* Having given informed consent
* Patient under a social security scheme
* Possibility to include a patient having already been included in the study but suffering from a new episode of hypercapnic non acidic Acute Respiratory Failure with a free interval of 3 months

Exclusion Criteria:

* Restrictive chronic neuromuscular or kyphoscoliotic respiratory insufficiencies
* Drug-induced Acute respiratory failure
* Pneumothorax (X-ray pulmonary detachment)
* Oxygen poisoning. In this case, PaCO2 will be asset again later with the purpose to include after oxygenotherapy decrease for a target SpO2 of 92% maximum
* Severe Acute Respiratory Syndrome (SARS) Coronavirus 2 (COVII) Pneumonia
* Tracheostomy
* Prior treatment with chronic or initiated NIV just prior to treatment (e.g. Intensive Care Unit)
* Respiratory Severity Criteria for Resuscitation Management
* Agitation or non-cooperation
* Pregnancy or breastfeeding
* Person participating in other biomedical research
* Any other reason that the investigator believes may interfere with the evaluation of the study objectives
* Person under judicial protection (guardianship, curatorship)
* Person deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Failure of the Nasal High Flow | Up to 2 weeks
  Failure of the Nasal High Flow is defined by the occurrence of respiratory acidosis (pH<7.35) within 2 weeks after admission

SECONDARY OUTCOMES:
Responding patients phenotype | At Day 30 after hospital discharge
  Phenotype will be characterized by the presence of one or more of the following elements : obesity hypoventilation syndrome, chronic obstructive pulmonary disease (COPD) emphysema, thoracic enlargement, bronchiectasis.
Etiology of acute respiratory failure | Up to 2 weeks
  The triggers of acute respiratory failure will be assessed : bacterial secondary infection, viral infection, bronchospasm, ...
Respiratory rate | Up to 2 weeks
  Respiratory rate will be recorded from Day 0 to Day 15, or until discharge (if less than 15 days).
Dyspnea | Up to 2 weeks
  Dyspnea will be assessed by the modified Borg scale rating of perceived exertion (RPE) from Day 0 to Day 15.
  The minimum value of the scale corresponding to no shortness of breath is 0 and the maximum value corresponding to dyspnea is 10. Higher score means a worse outcome.
pH | Up to 2 weeks
  pH will be assessed from Day 0 to Day 15.
Partial Pressure of Carbon dioxide (PCO2) | Up to 2 weeks
  PCO2 will be assessed from Day 0 to Day 15.
Bicarbonates | Up to 2 weeks
  HCO3- will be assessed from Day 0 to Day 15.
pCO2 normalization time | Up to 2 weeks
ROX index | Up to 2 weeks
  ROX index will be performed from Day 0 to Day 15.
Length of hospital stay | Up to 2 weeks
  Duration will be recorded in days medically necessary in the pneumology department
Comfort Visual Analogic Scale (VAS) | Up to 2 weeks
  Patient's comfort will be assessed on a Visual Analogic Scale at Day 0, Day 7 and Day 15 or at hospital discharge.
  The minimum value of the scale, corresponding to no discomfort is 0 and the maximum value corresponding to the maximum discomfort, is 10. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile MAINCENT, MD, Study Director — Centre Hospitalier Princesse Grace
Locations (3):
- France (2):
  - Centre Hospitalier de Cannes, Cannes, Alpes Maritime
  - Centre Hospitalier Intercommunal de Toulon- La Seyne sur Mer - Hôpital Sainte Musse, Toulon, Var
- Centre Hospitalier Princesse Grace, Monaco, Monaco